CLINICAL TRIAL: NCT05068258
Title: Lymphovenous Bypass (LVB) Promotes Healing Process of Venous Leg Ulcers
Brief Title: Lymphovenous Bypass Manage Venous Leg Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202105094RIND
Record Dates: First submitted 2021-09-06; First posted 2021-10-05 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-03

CONDITIONS: Venous Leg Ulcer; Lymphovenous Edema
Keywords: Chronic Venous Insufficiency; Lymphovenous Bypass
MeSH Terms: conditions — Varicose Ulcer | interventions — Drug Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Venous leg ulcers patients undergoing lymphovenous bypass (Experimental)
  Interventions: Procedure: Lymphovenous bypass, including lymphaticovenular anastomosis/implantation

INTERVENTIONS:
Procedure: Lymphovenous bypass, including lymphaticovenular anastomosis/implantation — Lymphovenous bypass (LVB) is a supermicrosurgical technique by diverting lymphatic drainage into venous system. Simultaneously, we performed LVB at ipsilateral foot dorsum and debride the VLUs and resurface the wound primarily or by skin graft depending on defect size.

SUMMARY:
Leg ulcers are areas of epidermal discontinuity in lower limbs with causes of venous, arterial, diabetic, pressure, traumatic, allergic, or inflammation. Chronic venous leg ulcers (VLUs) are defined as leg ulcers persisting for 4 weeks or more, a.k.a C6 in CEAP classification of chronic venous insufficiency (CVI) and account for up to 70% of all chronic leg ulcers exhibiting overall prevalence of up to 2% in the general population of western countries with significant morbidity and a negative socioeconomic impact. Wound care, debridement, bed rest with leg elevation, and compression are basic approaches for chronic VLUs. Meanwhile, numerous medical and surgical interventions were developed to promote wound healing and to prevent recurrence by focusing on pathophysiology of chronic VLUs. However, many strategies just have adjuvant effects or exert debatable benefits.

The lymphatic system been considered important for removal of excessive fluid from the interstitial space, absorption of fat from the intestine and the immune system, actively involved in regulation of immune cell trafficking and inflammation. Emerging lymphovenous bypass (LVB), a supermicrosurgical technique diverting lymphatic drainage into venous system in dealing with lymphedema, not only restores TH1 and TH2 imbalance, but decreases oxidative stress and increases antioxidant capacity in the serum of lymphedema patients. Clinically, LVB could be an alternative treatment option for patients with lymphorrhea.

Based on these facts, the investigators hypothesis that lymphatic hypertension and lymph impregnation contributes chronic venous leg ulcer formation and propose a novel strategy, using LVB to treat patients with refractory/recurrent chronic VLUs. The preliminary results revealed promising results and the investigators would go on clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20~80 years
* Gender: All
* Poor wound healing after standard wound management for 4 weeks
* Deep vein thrombosis (DVT) has been ruled out by Duplex and Computer tomography or DVT has been treated
* Wound care with nursing specialty
* Recognize and agree to join this trial

Exclusion Criteria:

* Autoimmune status, such as systemic lupus erythematosus
* Heart, lung, kidney or liver failure patients
* Radiation related wound or cancer wound
* Those who cannot understand the trial
* Age less than 20 years or elder than 80 years
* Pregnancy
* Those who was Risky to receive general anesthesia or surgery
* Allergy to Patent Blue V or Gentian Violet

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Healing process of venous leg ulcers | Postoperative 4~8 weeks
  Clinical assessment of wound healing in surface area (centimeter square)
Healing process of venous leg ulcers | Postoperative 12 weeks
  Clinical assessment of wound healing in surface area (centimeter square)
Healing process of venous leg ulcers | Postoperative 24 weeks
  Clinical assessment of wound healing in surface area (centimeter square)

SECONDARY OUTCOMES:
The venous leg ulcer quality of life (VLU-QoL) questionnaire (Chinese version verified), 0 (minimum) ~ 100 (maximum), higher scores mean a worse outcome | Preoperative
  The questionnaire evaluates 3 dimesions including activities, psychological and symptom distress aspect of patient having venous leg ulcers.
The venous leg ulcer quality of life (VLU-QoL) questionnaire (Chinese version verified), 0 (minimum) ~ 100 (maximum), higher scores mean a worse outcome | Postoperative 12 weeks
  The questionnaire evaluates 3 dimesions including activities, psychological and symptom distress aspect of patient having venous leg ulcers.
Venous Clinical Severity Score (VCSS), 0 (minimum) ~ 30 (maximum), higher scores mean a worse outcome | Postoperative 12 weeks
  Scoring system of chronic venous insufficiency

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Chuan Chao, MD, PhD, Study Director — National Taiwan University Hospital
Locations (1):
- Sung-Chuan Chao, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No